CLINICAL TRIAL: NCT06994273
Title: Analgesic and Sedative Effect of Fentanyl Versus Dexmedetomidine Infusion in Post-Operative Mechanically Ventilated Children After Open Abdominal Surgeries. Randomized Controlled Trial
Brief Title: Analgesic and Sedative Effect of Fentanyl Versus Dexmedetomidine Infusion in Post-Operative Mechanically Ventilated Children After Open Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Mohamed Abotaleb, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR315/8/23
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Analgesic; Sedative; Fentanyl; Dexmedetomidine; Infusion; Postoperative; Mechanical Ventilation; Children; Open Abdominal Surgeries
MeSH Terms: interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl group (Experimental): Patients received fentanyl as a 1 μg/kg bolus over 10 min, followed by a 1-5 μg/kg/hr intravenous infusion after 10-15 minutes
  Interventions: Drug: Fentanyl
- Dexmedetomidine group (Experimental): Patients received dexmedetomidine as a 1 μg/kg bolus over 10 min, followed by a 0.2-0.7 μg/kg/hr intravenous infusion after 10-15 minutes.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl — Patients received fentanyl as a 1 μg/kg bolus over 10 min, followed by a 1-5 μg/kg/hr intravenous infusion after 10-15 minutes.
  Arms: Fentanyl group
Drug: Dexmedetomidine — Patients received dexmedetomidine as a 1 μg/kg bolus over 10 min, followed by a 0.2-0.7 μg/kg/hr intravenous infusion after 10-15 minutes.
  Arms: Dexmedetomidine group

SUMMARY:
This study aimed to compare the efficacy and safety of fentanyl versus dexmedetomidine infusion in this population.

DETAILED DESCRIPTION:
Appropriate sedation and analgesia are essential components in the post-operative care of critically ill children in the pediatric intensive care unit (PICU), especially those who need mechanical ventilation.

Fentanyl is an opioid analgesic that is 50-100 times more potent than morphine. It is used frequently because of its ability to provide rapid analgesia. A single dose of fentanyl significantly reduced pain behaviors and changes in heart rate. It also increased the growth hormone level.

Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with significant sedative and analgesic effects. Some studies have investigated its role in adult and pediatric intensive care, as a primary sedative or a second line following failure of benzodiazepines or opioid sedation, as a bridge for extubation, for substance withdrawal, and to decrease intensive care unit (ICU) delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age from 4 to 11 years.
* Both sexes.
* Children who required a minimum of 24 hrs of mechanical ventilation following open abdominal surgeries

Exclusion Criteria:

* Patients with significant congenital anomalies.
* Chromosomal abnormalities.
* Neurologic conditions prohibiting sedation evaluation.
* Neuromuscular diseases.
* Those receiving neuromuscular blockers

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Weaning eligibility | 48 hours postoperatively
  The time from ventilator weaning eligibility was monitored until discharge.

SECONDARY OUTCOMES:
Time from eligibility to extubation | 60 min postoperatively
  Time from eligibility to extubation was monitored until discharge.
Mean arterial pressure | 48 hours post-infusion initiation
  Mean arterial pressure was continuously monitored and recorded at baseline and 2, 5, 10, 15, 30 minutes, 2, 6, 12, 24, and 48 hrs post-infusion initiation.
Heart rate | 48 hours post-infusion initiation
  Heart rate was continuously monitored and recorded at baseline and 2, 5, 10, 15, 30 minutes, 2, 6, 12, 24, and 48 hrs post-infusion initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Abotaleb AM, Elsheikh MR, Elshimy KM, AbdelFattah ME. Analgesic and Sedative Effect of Fentanyl Versus Dexmedetomidine Infusion in Postoperative Mechanically Ventilated Children After Open Abdominal Surgeries: Randomized Controlled Trial. Anesthesiol Res Pract. 2025 Jul 3;2025:9699738. doi: 10.1155/anrp/9699738. eCollection 2025. PMID 40642177